CLINICAL TRIAL: NCT00978133
Title: Prospective Randomized Study to Evaluate the Use of DERMABOND ProPen (2-octylcyanoacrylate) in the Closure of Abdominal Wounds Versus Closure With Skin Staples in Patients Undergoing Elective Colectomy.
Brief Title: Study of DERMABOND ProPen in Closure of Colectomy Wounds
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in accrual of study subjects, small numbers of potential subjects
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dermabond colectomy wounds
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Wound
Keywords: Colectomy; Closure; Wound; Dermabond; Propen
MeSH Terms: conditions — Wounds and Injuries | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Skin Staples (Active Comparator): Skin closure with skin staples
  Interventions: Procedure: Skin closure with skin staples
- Dermabond (Experimental): Closure of abdominal wound with dermabond (2-octylcyanoacrylate)
  Interventions: Procedure: Dermabond ProPen (2-octylcyanoacrylate)

INTERVENTIONS:
Procedure: Dermabond ProPen (2-octylcyanoacrylate) — Application of 2 layers of Dermabond to abdominal wounds after closure of deep layers
  Other Names: Dermabond ProPen
  Arms: Dermabond
Procedure: Skin closure with skin staples — Skin closure with skin staples
  Arms: Skin Staples

SUMMARY:
2-octylcyanoacrylate (2-OCA) has been used extensively in clinical practice in trauma, plastic surgery, orthopaedic surgery, emergency medicine and paediatrics. Most studies on 2-OCA to date have focused on closure of short wounds, and only one has included closure of abdominal wounds in the context of general surgery. Here, the investigators will look at the results of closure of abdominal wounds in patients undergoing elective colectomies with 2-OCA, which is commercially available to us, versus closure with skin staples, which is the current standard technique of skin closure employed in the Department of Colorectal Surgery, Singapore General Hospital. The primary objective was to measure effectiveness of 2-OCA in 2 respects - the adequacy of wound healing and cosmesis, and the incidence of superficial wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective colectomies for benign or malignant conditions
* Midline vertical incisions or skin crease incisions
* Above the age of 21 years old
* Able to make own valid informed decisions

Exclusion Criteria:

* Patients undergoing surgery for recurrent or metastatic disease
* Surgery for surgical emergencies such as acute abdomen or bleeding
* Known allergy to DERMABOND ProPen Tissue Adhesive or any of its constituents (cyanoacrylate or formaldehyde)
* Patients on immunosuppression

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Wound healing | 3 months
Patient satisfaction | 3 months

SECONDARY OUTCOMES:
Superficial surgical site infections | 3 months
Time taken for wound closure | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Julian KP Ong, FRCSEd, Principal Investigator — Singapore General Hospital; Kok-Sun Ho, FRCS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Quinn J, Wells G, Sutcliffe T, Jarmuske M, Maw J, Stiell I, Johns P. Tissue adhesive versus suture wound repair at 1 year: randomized clinical trial correlating early, 3-month, and 1-year cosmetic outcome. Ann Emerg Med. 1998 Dec;32(6):645-9. doi: 10.1016/s0196-0644(98)70061-7. PMID 9832658
- [Background] Blondeel PN, Murphy JW, Debrosse D, Nix JC 3rd, Puls LE, Theodore N, Coulthard P. Closure of long surgical incisions with a new formulation of 2-octylcyanoacrylate tissue adhesive versus commercially available methods. Am J Surg. 2004 Sep;188(3):307-13. doi: 10.1016/j.amjsurg.2004.04.006. PMID 15450839